CLINICAL TRIAL: NCT05809141
Title: Comparison Between Thromboelastography and Conventional Coagulation Tests in Pediatrics With Chronic Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennat-Allah Hesham Abdelraheem, resident doctor of pediatrics department, Assiut University
Other Study IDs: thromboelastography
Record Dates: First submitted 2023-03-18; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Thromboelastography; Conventional Coagulation Tests; Chronic Liver Disease
MeSH Terms: interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: thromboelastography — Thromboelastography (TEG), a whole blood viscoelastic test. TEG detects the clotting time, clotting kinetics and clot stability to more comprehensively evaluate haemostatic status by several parameters, mainly including reactive time (R), kinetic time (K), angle (α), maximum amplitude (MA) and lysis-30 .

SUMMARY:
* Compare between thromboelastography (TEG) and conventional coagulation tests (CCT) in children with chronic liver disease who admitted to Assiut University Children Hospital.
* Detect the advantages of TEG in predicting the risk of bleeding, assessing haemostasis and guiding blood product transfusion for each coagulation defect .

DETAILED DESCRIPTION:
The liver is the largest solid organ in the body with a mass of 1200-1500 g. It develops embryologically as a glandular outgrowth of the primitive gut, forming also the largest gland of the body . The liver is the major site of synthesis of haemostatic factors and clearance of activated haemostatic factors . These factors are important to maintain dynamic balance of physiological haemostasis, including primary haemostasis (i.e. interaction between platelet [PLT] and vessel wall), coagulation cascade and fibrinolysis . Consequently, in patients with liver dysfunction, a complicated disorder of haemostatic system arises, causing both bleeding and thromboembolic complications .

Chronic liver disease (CLD) is a progressive deterioration of liver functions for more than six months, which includes synthesis of clotting factors, other proteins, detoxification of harmful products of metabolism, and excretion of bile . The spectrum of etiologies is broad for chronic liver disease, which includes toxins, alcohol abuse for a prolonged time, infection, autoimmune diseases, genetic and metabolic disorders . The common causes for chronic liver disease (CLD) in children are hepatitis B, hepatitis C, hepatitis D, autoimmune hepatitis and metabolic disorders like Wilson's disease and α-1 antitrypsin deficiency . In majority of the patients the etiology remains uncertain. Signs and symptoms of CLD can be nonspecific, such as fatigue, anorexia, weight loss, or depend upon the complication that the patient has developed. The three significant complications are because of portal hypertension (esophageal varices, ascites), hepatocellular insufficiency (e.g., jaundice, hepatic encephalopathy), and hepatocellular carcinoma .

Among complications of chronic liver disease: variceal bleeding, ascites, spontaneous bacterial peritonitis (SBP), hepatic encephalopathy, hepatorenal syndrome, hepatopulmonary syndrome and hepatocellular carcinoma (HCC) .

There are various scoring systems used to assess the severity of chronic liver disease .

Physiological haemostasis includes primary haemostasis, coagulation cascade and fibrinolysis, which are involved with various haemostatic factors. Haemostatic tests mainly include conventional coagulation tests (CCTs) and thromboelastography (TEG) test. CCTs mainly includes PLT count, PT, APTT, and fibrinogen (FIB), d-dimer and fibrinogen degradation products (FDP) concentrations. PLT count reflects primary haemostasis by quantitative assessment of PLT. PT and APTT reflect coagulation cascade by assessment of pro-coagulants involved in the extrinsic and intrinsic pathways, respectively. FIB concentration reflects coagulation cascade by quantitative assessment of FIB. D-dimer and FDP concentrations reflect fibrinolytic activity by quantitative assessment of d-dimer and FDP .

Thromboelastography (TEG), a whole blood viscoelastic test. TEG detects the clotting time, clotting kinetics and clot stability to more comprehensively evaluate haemostatic status by several parameters, mainly including reactive time (R), kinetic time (K), angle (α), maximum amplitude (MA) and lysis-30 . R reflects the activity of coagulation factors by detecting the time of fibrin formation. K and α reflect the fibrinogen function by detecting the rate of clot development. MA reflects the platelet function by detecting the maximum clot strength. Lysis 30 reflects fibrinolytic activity by detecting the degree of fibrinolysis .

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic liver disease of any aetiology as (congenital hepatic fibrosis, liver cirrhosis, autoimmune hepatitis, Wilson disease, metabolic liver disease and others ).
* Patients aged 6m- 18y .

Exclusion Criteria:

* Patients who received transfusion of blood products within 48hr prior to sample collection.
* Patients who are on therapy with antiplatelet drugs or anticoagulants.
* Patients with history of primary disease with coagulation disturbance (paroxysmal nocturnal hemoglobinuria, polycythemia, idiopathic thrombocytopenia, haemophilia.
* Patients with concomitant chronic kidney disease.

Ages: 6 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients aged 6m-18y with chronic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Detect the clotting time, clotting kinetics and clot stability | Baseline
  By thromboelastography parameters
compare between thromboelastography and conventional coagulation tests | Baseline
  in evaluation of haemostatic status in pediatrics with chronic liver disease .
Detect the advantages of thromboelastography | Baseline
  predicting the risk of bleeding, assessing haemostasis and guiding blood product transfusion for each coagulation defect .

REFERENCES:
- [Background] Yang LL. Anatomy and Physiology of the Liver. Anesthesia for Hepatico-Pancreatic-Biliary Surgery and Transplantation. 2021:15-40.
- [Background] Amitrano L, Guardascione MA, Brancaccio V, Balzano A. Coagulation disorders in liver disease. Semin Liver Dis. 2002 Feb;22(1):83-96. doi: 10.1055/s-2002-23205. PMID 11928081
- [Background] Versteeg HH, Heemskerk JW, Levi M, Reitsma PH. New fundamentals in hemostasis. Physiol Rev. 2013 Jan;93(1):327-58. doi: 10.1152/physrev.00016.2011. PMID 23303912
- [Background] He Y, Yao H, Ageno W, Mendez-Sanchez N, Guo X, Qi X. Review article: thromboelastography in liver diseases. Aliment Pharmacol Ther. 2022 Aug;56(4):580-591. doi: 10.1111/apt.17080. Epub 2022 Jun 14. PMID 35698893
- [Background] Sharma A, Nagalli S. Chronic Liver Disease. 2023 Jul 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554597/ PMID 32119484
- [Background] Chronic hepatitis and autoimmune chronic active hepatitis. In: Alex P.Movat (eds). Liver disorders in childhood 3rd edition. Oxford, Butterworth- Heinemann Ltd, 1994, pp. 180-96.
- [Background] Viral hepatitis/Chronic hepatitis/Portal hypertension. In: Sherlock S, Dooley J, (eds). Diseases of liver and biliary system 10th edition. Oxford, Blackwell Science Ltd, 1997, pp. 162-3, 265-333.
- [Background] Janko N, Majeed A, Kemp W, Roberts SK. Viscoelastic Tests as Point-of-Care Tests in the Assessment and Management of Bleeding and Thrombosis in Liver Disease. Semin Thromb Hemost. 2020 Sep;46(6):704-715. doi: 10.1055/s-0040-1715475. Epub 2020 Sep 15. PMID 32932542